CLINICAL TRIAL: NCT05010499
Title: Hip Arthroscopy; Femoral Nerve Block or Fascia Iliaca Block: A Randomized Control Trial
Brief Title: Hip Arthroscopy; Femoral Nerve Block or Fascia Iliaca Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maha sadek El Derh, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 143/2021
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Anlgesia for Hip Arthroscopy by Assessing Quality of Different Type of Regional Block, Femoral Nerve Block Versus Fascia Iliaca Block
MeSH Terms: interventions — Levobupivacaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: patients undergoing hip arthroscope are divided into 2 groups. patients either receive femoral nerve block or fascia iliaca block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: neither the patients nor the treating doctor know the type of block patient received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral nerve block (Active Comparator): Patients will receive femoral nerve block (20 ml levobupivacaine 0.25%) after general anesthesia for hip arthroscpe
  Interventions: Drug: Levobupivacaine
- Fascia iliaca block (Active Comparator): Patients will receive fascia iliaca block (40 ml levobupivacaine 0.25%) after general anesthesia for hip arthroscpe
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — femoral nerve block receives 20 ml of levobupivacaine 0.25%
  Other Names: Bupivacaine hydrochloride (Marcaine)
  Arms: Femoral nerve block
Drug: Levobupivacaine — Fascia iliaca block receives 40 ml of levobupivacaine 0.25%
  Other Names: Bupivacaine Hydrochloride (Marcaine)
  Arms: Fascia iliaca block

SUMMARY:
Patients undergoing hip arthroscopy will be divided into 2 groups after receiving general anesthesia. 1 group will receive femoral nerve block and the other one will receive fascia iliaca block. Postoperative total rescue analgesia will recorded in both groups, and in which group early ambulation will take place .

DETAILED DESCRIPTION:
Patients undergoing hip arthaoscope will be conducted to operating room, where standard intraoperative monitoring will be applied, pulse oximetry, 5 lead ECG then peripheral cannulation. Anesthesia will be induced with fentanyl 1.5μg/kg, midazolam 0.1-0.5 mg/kg, cis-atracurium 0.15 mg/kg followed by intubation. Then anesthesia will be maintained with isoflurane1-1.5% Patients will be divided into two groups according to the randomization envelopes:

Group (A) :( 15 patients) the fascia iliaca block: Patient in the supine position, skin will be disinfected and linear transducer (8-12 MHZ) will be positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer will be moved laterally until the sartorius muscle is identified. Echogenic needle (Bajunk, 80 m.m length) will be inserted in-plane, as it will pass through fascia iliaca, the fascia will be first seen indented by the needle. While piercing the fascia, a "pop" may be felt, and the fascia may be seen to "snap" back on the US image (SONOSITE). After negative aspiration, 1-2 mL of local anesthetic is injected to confirm the proper injection plane between the fascia and the iliopsoas muscle. A proper injection will result in the separation of the fascia iliaca by the local anesthetic in the medial-lateral direction from the point of injection as described. Releasing the pressure of the transducer may reduce the resistance to injection and improve the distribution of local anesthetic. If the spread is deemed inadequate, additional injections laterally or medially to the original needle insertion or injection can be made to facilitate the medial-lateral spread (the injection is stopped and the needle repositioned before continuing. Additional injections may be made to ensure adequate spread) (Yun MJ, et al., 2009). 40 mL of 0.25% levobupivacaine will be given. The success of the nerve block is best predicted by documenting the spread of local anesthetic toward the femoral nerve medially and underneath the sartorius muscle laterally (L. Hanna, et al., 2014).

Group (B): Control group, (15 patients) femoral nerve block: With the patient in the supine position, the skin over the femoral crease will be disinfected and the transducer will be positioned to identify the femoral artery and nerve. If the nerve is not immediately apparent lateral to the artery, tilting the transducer proximally or distally often helps to image and highlight the nerve from the iliacus muscle and the more superficial adipose tissue. Once the femoral nerve is identified, the needle will be inserted in-plane in a lateral to medial orientation and advanced toward the femoral nerve (Mariano E.R ,et al., 2013). Once the needle tip is adjacent (either above, below, or lateral) to the nerve, and after careful aspiration, 1-2 mL of local anesthetic will be injected to confirm proper needle placement that will push the femoral nerve away from the injection followed by total volume of 20 ml 0.25% levobupivacaine (Lamaroon A. et al., 2014) The blocks will be performed by the expert anesthesia staff, and then positioning of patients will be done for the hip arthroscopy. Another blinded doctor to the type of block received will attend the surgery and manage and record any additional intraoperative analgesic requirements.

Postoperatively, timing for the first rescue analgesia will be recorded, if VAS is more than 5, 25 mg pethidine will be given. If no improvement second rescue analgesia in form 5 mg morphine will be given .Also total narcotics demand will be recorded with measurement of (VAS) hourly in the first 4 hours postoperatively then every 4 hours for 8 hours .Early ambulation will be assessed and recorded together with assessing the weakness of quadriceps femoris.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 45 years ,ASA I and II undergoing hip arthroscope.

Exclusion Criteria:

* Age less than 21 or more than 45 years
* ASA IV
* Those who have an emergency surgery, or patients scheduled for complicated surgeries
* Those who have a history of allergy to levobupivacaine
* local skin site infections.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Record the time patients require analgesia postoperatively | 12 hours
  Assessment of postoperative pain score by Visual analogue Scale (VAS) and the time of demand for first rescue analgesia

SECONDARY OUTCOMES:
postoperative ability to ambulate. | 24 hours postoperative
  Assess the time patients start to ambulate postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- maha sadek El Derh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided